CLINICAL TRIAL: NCT06321991
Title: Nodular Shrinking in Stage 0 Dupuytren Disease: an Evidence-based Approach for Early Stage Treatment to Prevent Progression to Advanced Finger Contractures
Brief Title: Nodular Shrinking in Dupuytren Disease
Acronym: Echo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S68382
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Intervention Model Description: Simple random allocation will be ensured by the principal investigators' designated staff (study nurse of IORT), who will not be involved in recruiting trial participants, medical care, drug administration or follow-up, through the generation of a random numbers table with computer software program. A randomization list will be prepared by the Sponsor's designated staff, not involved in recruiting Trial participants, medical care, drug administration or follow-up.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To avoid bias, treatment arms will be blinded to Investigators, Trial staff, participants,.. as follows: vitamin E creme will be packaged and labelled in such a way that the visual appearance, nor the smell and/or touch of the creme can be distinguished from placebo (Vaseline).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupuytren Disease patients receiving Vasiline (Placebo) (Placebo Comparator): 40 patients with Dupuytren Disease (primary DD nodules: stage 0, no contracture in the involved hand) will be randomized into the group where they will receive Vasiline
  Interventions: Drug: Vitamin E-creme (Remederm®) vs Vaseline (Placebo); Procedure: Ultrasound measurement
- Dupuytren Disease patients receiving Remederm® (Vitamine E creme) (Active Comparator): 40 patients with Dupuytren Disease (primary DD nodules: stage 0, no contracture in the involved hand) will be randomized into the group where they will receive Remederm® (Vitamine E creme)
  Interventions: Drug: Vitamin E-creme (Remederm®) vs Vaseline (Placebo); Procedure: Ultrasound measurement

INTERVENTIONS:
Drug: Vitamin E-creme (Remederm®) vs Vaseline (Placebo) — Louis Widmer Remederm® Face Cream Without Perfume 50 ml is a skin care product that contains vitamin E as an active ingredient. Before applying Remederm®, the following are advised: On dry clean skin thoroughly before applying Remederm®, apply a layer of cream cutaneous to the hand palm, twice a day: morning and evening, massage cream into skin until absorbed. This procedure is applied by the patient treated with Vaseline or Remederm®.
Procedure: Ultrasound measurement — Nodule evolution will be measured with ultrasound.

SUMMARY:
Dupuytren disease (DD) is a common hand disorder with disabling finger contractures that may require surgery to restore function. In the early stages of the disease, the nodules (Tubiana stage 0) are usually painless, but a reason for concern to many patients. Not rarely, lifestyle measures and even risky treatment options as radiotherapy are advised, yet no therapy to prevent disease evolution has a solid proven effect. Furthermore, reliable non-invasive measurement of early stage DD is not validated.

Evidence was found that pharmacotherapy may influence DD evolution, but valuable clinical trials are limited. Case series and non-published explorative follow-up suggested local treatment with antioxidant vitamin E to possibly interfere with an evolution of DD nodules to contracting strands. This study aims to provide evidence on efficiency of this non-invasive treatment option.

Secure measurement of nodule evolution is a clinical challenge. To measure this evolution, ultrasound and MRI scanning are currently being performed. Stage 0 (nodules) is more challenging to quantify. A strict individual follow-up by the treating clinician is needed to standardize measurement of selected (treated) nodules. Therefore, simple ultrasound by the treating clinician may provide an good tool to collect data. This study aims to introduce and validate this non-invasive scan method and provide a prospective double blind investigation of a measurable effect of non-invasive preventive treatment for stage 0 DD to improve clinical outcome.

DETAILED DESCRIPTION:
Dupuytren disease (DD) is a common hand disorder with disabling finger contractures that may require surgery to restore function. The contractures are caused by progressive fibroproliferative tissue forming nodules and strands in the palmar fascia that eventually cause loss of finger extension. In the early stages of the disease, the nodules (Tubiana stage 0) are usually painless, but a reason for concern to many patients. They often seek the hand surgeon's advice and worry about losing hand function the coming years, commonly requesting for precautionary measures to stop evolution towards contractures (Tubiana stage 1-4). Not rarely, lifestyle measures and even risky treatment options as radiotherapy are advised, yet no therapy to prevent disease evolution has a solid proven effect. Furthermore, reliable non-invasive measurement of early stage DD is not validated.

However, this is needed to explore any efficient preventive treatment that may be cost-efficient for patients and healthcare.

Evidence was found that pharmacotherapy may influence DD evolution, but valuable clinical trials are limited. Case series and non-published explorative follow-up suggested local treatment with antioxidant vitamin E to possibly interfere with an evolution of DD nodules to contracting strands. Therefore, it is recommended to consider local creams to the palms in such situation.

This study aims to provide evidence on efficiency of this non-invasive treatment option. Secure measurement of nodule evolution is a clinical challenge. To measure this evolution, ultrasound and MRI scanning are currently being performed. In clinical practice, although clinical staging of contractures is reliable, stage 0 (nodules) is more challenging to quantify. If observed, nodules (evolution) are often measured by clinical yardstick assessment. However, this technique is unvalidated and unreliable with inevitable significant inter- and intra-observer unreliability, which may improve with sonography. A strict individual follow-up by the treating clinician is needed to standardize measurement of selected (treated) nodules. Therefore, simple ultrasound by the treating clinician may provide an good tool to collect data. The V-Scan (simple office-based Bluetooth ultrasonography) may aid to achieve this and its use is successfully implemented since 1 year at the hand Surgery department at Université Catholique de Louvain (UCL) by and under supervision of Prof Dr X. Libouton.

This study aims to introduce and validate this non-invasive scan method and provide a prospective double blind investigation of a measurable effect of non-invasive preventive treatment for stage 0 DD to improve clinical outcome.

Rationale: Application of antioxidant creme cause V-scan measurable arrest or even shrinking of the nodules in stage 0 of DD.

ELIGIBILITY:
Inclusion Criteria:

* The participant or his/her legally authorized representative voluntary signed the informed consent prior to the first assessment.
* Participants are ≥ 18 years and diagnosed with primary Dupuytren disease.
* Included patients have a stage 0 DD (nodule of at least 5 mm in the involved hand without contracture).
* The participant has well distinguished noduli that are clearly visible on US (ultrasound)

Exclusion Criteria:

* Patients < 18 years.
* Patient included in an interventional trial with an investigational medicinal product.
* Patients with cognitive impairments, severe rheumatic disease and neurological disorders leading to flexion deformities of the fingers.
* Patients with prior Dupuytren surgery in the involved hand.
* Patients with a higher Tubiana grading than nodular stage 0.
* Open wound in the palm of the treated hand.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Downsizing of the largest nodule diameter | 1 year
  A significant downsize (>1mm because V-scan (ultrasonography) is accurate to 1mm) of the largest nodule diameter in the palm of the hand.

SECONDARY OUTCOMES:
VAS questionnaire on pain | 1 year
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). The patient is asked to rate their current level of pain by placing a mark on the line.
VAS questionnaire on satisfaction | 1 year
  The Visual Analogue Scale (VAS) measures satisfaction. The VAS consists of a 10cm line, with two end points representing 0 ('complete dissatisfaction') and 10 ('full satisfaction'). The patient is asked to rate their current level of satisfaction by placing a mark on the line.
QUICK Dash for functionality | 1 year
  This questionnaire asks the patient about the symptoms as well as the ability to perform certain activities. It consists of 11 items ranging from 1 ('not at all/no difficulty') to 5 ('extremely/unable').
Abe Diathesis scoring | Baseline
  An objective method to evaluate the risk of recurrence and extension of Dupuytren's disease. This scoring counts 1 point for each for bilateral, small finger surgery and if onset < 50 y. The scoring counts 2 points each for Ledderhose, knuckle pads, thumb / index disease. Diathesis score = sum of points. Increased risk for score > 4.
Range of motion | 1 year
  By using goniometry of Distal interphalangeal, Proximal Interphalangeal and metacarpophalangeal joints
Recurrence rate | 1 year
  Recurrence is defined as the clinical re-appearance of the treated nodules or a significant increase of diameter (>1mm) or evolution to a higher stage (Tubiana stage 1-4) of the disease than 0 at intake.

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Degreef, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No